CLINICAL TRIAL: NCT04284384
Title: Modifiable Risk Factors and Dementia - A Study Examining the Association Between Hearing Impairment in Mid-life and Cognitive Impairment in the HUNT4 70+ Study
Brief Title: Hearing Impairment as a Risk Factor for Dementia in Older Adults
Status: Completed | Type: Observational
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: Norwegian University of Science and Technology (Other); The Nord-Trøndelag Health Study (Unknown); The Norwegian Institute of Public Health (Unknown); University College London Hospitals (Other); University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 181009
Record Dates: First submitted 2020-02-06; First posted 2020-02-25 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Dementia; Hearing Loss
MeSH Terms: conditions — Dementia; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HUNT4 70+: All inhabitants of Nord-Trøndelag 70 years of age or older were invited to participate in HUNT4 70+.
- HUNT Trondheim 70+: All inhabitants of one district in Trondheim 70 years of age or older were invited to participate in HUNT4 70+.

SUMMARY:
This Doctor of Philosophy (PhD) project is part of a larger project on potentially modifiable risk factors for dementia in a life course perspective, with an overarching aim to improve prevention of dementia and thereby potentially relieve patient and caregiver distress and decrease societal load. The present PhD project will concentrate on confirming knowledge of HI as an independent risk factor for dementia and exploring potentially causative factors to explain this relationship.

DETAILED DESCRIPTION:
Despite a huge increase in the knowledge about disease mechanisms in various types of dementia in recent years, no curative treatment exists at present. Results from research on disease-modifying agents have been disappointing. This has led to an increased interest in other ways to reduce the prevalence of dementia. A recent report estimated that up to one third of dementia cases could be delayed or prevented by interventions directed at the most common risk factors. In the "Lancet commission on dementia prevention, treatment, and care", hearing impairment (HI) was identified as the potentially most important modifiable risk factor. Even though HI is considered an important modifiable risk factor, the evidence regarding the association between HI and dementia risk is still limited.

ELIGIBILITY:
Inclusion Criteria:

* Living in designated area

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: HUNT2 and HUNT4 hearing studies: Participants from 17 of the 24 municipalities in the county were offered and accepted a hearing examination, consisting of pure-tone audiometry and two questionnaires on hearing issues, such as use of hearing aids, noise exposure, and tinnitus.
  HUNT4 70+/HUNT Trondheim 70+: All participants 70 years of age or older are invited to participate in HUNT4 70+ including cognitive screening examinations.
Sampling Method: Non-Probability Sample
Enrollment: 6952 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Rate of dementia diagnosis in the HUNT 70+ study | 2017-2019
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5).
Rate of Minimal Cognitive Impairment (MCI) in the HUNT 70+ study | 2017-2019
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria DSM-5.
Rate of cognitive impairment defined as age- and education-adjusted thresholds on cognitive assessments scales | 2017-2019
  The participants have been assessed with the Montreal Cognitive Assessment scale and the ten-word recall test

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbæk, PhD, Principal Investigator — Norwegian Centre for Ageing and Health
Locations (1):
- Norwegian National Advisory Unit of Ageing and Health, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GjOra L, Strand BH, Bergh S, Borza T, Braekhus A, Engedal K, Johannessen A, Kvello-Alme M, Krokstad S, Livingston G, Matthews FE, Myrstad C, Skjellegrind H, Thingstad P, Aakhus E, Aam S, Selbaek G. Current and Future Prevalence Estimates of Mild Cognitive Impairment, Dementia, and Its Subtypes in a Population-Based Sample of People 70 Years and Older in Norway: The HUNT Study. J Alzheimers Dis. 2021;79(3):1213-1226. doi: 10.3233/JAD-201275. PMID 33427745
- [Derived] Myrstad C, Engdahl BL, Costafreda SG, Krokstad S, Livingston G, Selbaek G. Hearing and cognitive scores measured with the Montreal Cognitive Assessment Scale in The HUNT Study, Norway. Alzheimers Dement. 2025 Feb;21(2):e14514. doi: 10.1002/alz.14514. Epub 2025 Jan 23. PMID 39846386
- [Derived] Myrstad C, Engdahl BL, Costafreda SG, Krokstad S, Lin F, Livingston G, Strand BH, Ohre B, Selbaek G. Hearing impairment and risk of dementia in The HUNT Study (HUNT4 70+): a Norwegian cohort study. EClinicalMedicine. 2023 Dec 4;66:102319. doi: 10.1016/j.eclinm.2023.102319. eCollection 2023 Dec. PMID 38192588

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT04284384/SAP_000.pdf